CLINICAL TRIAL: NCT02901522
Title: Tele-spirometry in Primary Care - Randomized Clinical Trial Cluster: the Effectiveness of Multifaceted Intervention in Symptoms Patients With Respiratory Illness.
Brief Title: Tele-spirometry in Primary Care - Randomized Clinical Trial Cluster: the Effectiveness of Telemedicine in Asthma
Acronym: RESPIRANET-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Prefeitura Municipal de Porto Alegre (Unknown); Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 227190 Asthma
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
Keywords: telemedicine; asthma control test; Primary Health care; spirometry
MeSH Terms: conditions — Asthma | interventions — BaseLine dental cement; Remote Consultation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Spirometry (baseline) Spirometry (20 - 22weeks)
  Interventions: Other: Spirometry (baseline); Other: Spirometry (20 - 22weeks)
- Telemedicine (Experimental): Spirometry (baseline) Telemonitoring Teleconsultation Spirometry (20 - 22weeks)
  Interventions: Other: telemonitoring; Other: Spirometry (baseline); Other: Spirometry (20 - 22weeks); Other: Teleconsultation

INTERVENTIONS:
Other: telemonitoring — Patients is evaluated by telemonitoring (phone call nurse - 45 and 90 days).
  Arms: Telemedicine
Other: Spirometry (baseline) — Patients is evaluated by Asthma Control Test and spirometry at baseline and after 20 weeks.
Other: Spirometry (20 - 22weeks) — Patients is evaluated by Asthma Control Test and spirometry at baseline and after 20 weeks.
Other: Teleconsultation — The general practioner received phone call to asthma care.
  Arms: Telemedicine

SUMMARY:
The purpose of this study is to determine the effectiveness of telemedicine multifaceted intervention in symptoms patients with asthma.

DETAILED DESCRIPTION:
This study is a randomized clinical trial for patients with asthma from a primary care. The purpose is to determine the effectiveness of telemedicine (teleconsultation and telemonitoring) in control of asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* individual with diagnosis asthma, Asthma Control Test <20, spirometry from TelessaudeRS-Universidade Federal do Rio Grande do Sul (from randomization cluster)

Exclusion Criteria:

-low quality spirometries (inadequate)

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms control | 20 to 22 weeks
  Asthma Control Test (difference three points in the questionnaire ACT)

SECONDARY OUTCOMES:
Spirometry FVC | 20 to 22 weeks
  Spirometry parameters - FVC (forced vital capacity)
Spirometry FEV1 | 20 to 22 weeks
  Spirometry parameters - FEV 1 (forced expiratory volume in one second)

CONTACTS AND LOCATIONS:
Overall Officials: Erno Harzheim, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- TelessaudeRS-Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided